CLINICAL TRIAL: NCT04476550
Title: Developing a Potential Cure for Pompe Disease: Clinical Specimen Collection From Individuals With Pompe Disease
Brief Title: Clinical Specimen Collection From Pompe Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Serhat Gumrukcu, MD PhD (Other)
Collaborators: Frida Therapeutics LLC (Unknown)
Responsible Party: Sponsor-Investigator, Serhat Gumrukcu, MD PhD, Sponsor-Investigator, Seraph Research Institute
Organization: Seraph Research Institute (Other)
Other Study IDs: SRPH-LP-02/PoD
Record Dates: First submitted 2020-02-26; First posted 2020-07-20 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pompe Disease
Keywords: Pompe; Pompe Disease; HSPC; modified bone marrow stem cell
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mononuclear cells with GAA gene mutation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Filgrastim — 5 days of daily sub-cutaneous administration of 10mcg/kg filgrastim
  Other Names: Granulocyte-Colony Stimulating Factor (G-CSF)

SUMMARY:
Clinical specimens are required from individuals with Pompe Disease to support process and analytical development for a genetically modified autologous bone marrow cell product currently in preclinical research, FTX-PD01. The intent is for this product to be investigated in a subsequent clinical trial under a future FDA IND to treat Pompe Disease. Enrolled participants provide a venous blood specimen (approximately 20mL) to be used in preclinical studies and research and development of FTX-PD01. Subjects may eventually be asked to undergo mobilized leukapheresis for bone marrow stem cell collection and their specimens will be used to further develop the FTX-PD01 cell product, including a cGMP compliant process to be applied under the future FDA IND.

DETAILED DESCRIPTION:
This protocol is to collect blood and HSPC specimens from individuals with Pompe Disease. The first blood draw will be done at the first study visit and if eligible, the second collection will be done via mobilized leukapheresis at the second visit. The mobilized leukapheresis procedures will follow the facility's standard operating procedures and protocol requirements for mobilized leukapheresis.

Donors will be males or females between and including the ages of 3 years and 30 years. Volunteers will provide written informed consent and meet all inclusion and exclusion criteria. Each participant can be in the study for up to 120 days (3 months).

The study will be conducted in accordance with human research for the purposes of obtaining clinical specimens for research. There is no endpoint for this study, however, data collected from this study will include, but not be limited to, gender, demographics, medical history, clinical laboratory values, and volume of the blood collected. The data will be summarized in future studies reporting results from a future clinical trial under FDA IND.

ELIGIBILITY:
Inclusion Criteria:

* Male of female aged 3-30
* Documented diagnosis of Pompe Disease
* Participants who has not participated in a cell or gene therapy trial for Pompe Disease

Exclusion Criteria:

* Active acute infection at screening
* Uncontrolled diabetes
* Uncontrolled hypertension
* Active DIC, bleeding or coagulopathy which cannot be corrected with minimal intervention
* Symptomatic, uncontrolled or severe intercurrent illness that would compromise the ability to tolerate blood collection or mobilized leukapheresis procedure
* Systemic chemotherapy less than or equal to 2 weeks (6 weeks for clofarabine or nitrosoureas) or radiation therapy less than or equal to 3 weeks prior to leukapheresis
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test at screening
* Any patient that in the opinion of the investigator is not medically stable to undergo the leukapheresis procedure or will not comply with the visit schedules or procedures

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Otherwise healthy individuals diagnosed with Pompe Disease.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Collection of blood | Up to 20 days
  Collection of peripheral blood (up to 20ml)

SECONDARY OUTCOMES:
Collection of HSPCs | Up to 100 days
  Collection of HSPCs through G-CSF mobilized leukapheresis

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Gumrukcu, MD PhD, Principal Investigator — Seraph Research Institute
Locations (1):
- Seraph Research Institute, Toluca Lake, California, United States

IPD SHARING:
Plan to Share IPD: No